CLINICAL TRIAL: NCT00658606
Title: Efficacy and Safety of Alefacept in Combination With Narrow-band UVB (nbUVB) Compared to Alefacept Alone in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Assess the Efficacy and Safety of Alefacept With Narrow Band Ultraviolet B Phototherapy (nbUVB) vs. Alefacept Alone in Chronic Plaque Psoriasis Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AME-001
Record Dates: First submitted 2008-04-10; First posted 2008-04-15 (Estimated); Results first posted 2011-04-22 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Plaque Psoriasis
Keywords: plaque psoriasis; alefacept; Amevive; narrow band ultraviolet B; phototherapy
MeSH Terms: interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alefacept alone (Active Comparator): 15 mg alefacept intramuscularly (IM) once weekly for 12 weeks
  Interventions: Drug: alefacept
- Alefacept + nbUVB (Experimental): 15 mg alefacept intramuscularly once weekly and narrow band Ultraviolet B (nbUVB) phototherapy 3 times per week for 12 weeks
  Interventions: Procedure: Narrow Band UVB Phototherapy

INTERVENTIONS:
Drug: alefacept — IM
  Other Names: Amevive; ASP0485
  Arms: Alefacept alone
Procedure: Narrow Band UVB Phototherapy — UVB Phototherapy
  Arms: Alefacept + nbUVB

SUMMARY:
Assess the efficacy and safety of alefacept with nbUVB compared to alefacept alone in chronic plaque psoriasis subjects. Combination therapy may improve the clinical response to psoriatic subjects as both modalities have an effect on T cells

ELIGIBILITY:
Inclusion Criteria:

* Subject has given written informed consent
* Subject has a diagnosis of moderate to severe chronic plaque psoriasis involving >=10% with a Psoriasis Area and Severity Index (PASI) score >=10 at Baseline
* Subject has CD4+ T lymphocyte (CD4) count at or above the lower limit of normal
* Male and female subjects must use an adequate means of contraception from screening to end of study.

Exclusion Criteria:

* Subject who received alefacept in the past
* Subject who has shown no improvement following an adequate course of nbUVB in the past
* Subject who has been treated in the past with either therapy or cyclosporine
* Subject with any active cancer, including skin cancer at Baseline
* Subject with erythrodermic, pustular or predominantly guttate psoriasis
* Subject who has used treatment for psoriasis prior to Baseline as follows:

  * Topical treatment within 14 days
  * Oral treatment within 28 days
  * Broad band UVB (bbUVB) or nbUVB treatment within 56 days
  * Biological treatment within 84 days
* Serious local infection or serious systemic infection within the 3 months prior to the first dose of study drug
* Subject with a history of drug or alcohol abuse within the past 2 years
* Subject that is known to be infected with the AIDS virus
* Subject with any other skin disease or other disease that might interfere with psoriasis status assessments
* Female subject who is nursing, pregnant or planning to become pregnant while in this study
* Subject who is currently enrolled in any other investigational drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Canada, Inc.
Locations (11):
- Canada (11):
  - Calgary, Alberta
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - St. John's, Newfoundland and Labrador
  - London, Ontario
  - Markham, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sainte-Foy, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Background] Lui H, Gulliver W, Tan J, Hong CH, Hull P, Shear NH, Paradiso-Hardy F, Bissonette R. A randomized controlled study of combination therapy with alefacept and narrow band UVB phototherapy (UVB) for moderate to severe psoriasis: efficacy, onset, and duration of response. J Drugs Dermatol. 2012 Aug;11(8):929-37. PMID 22859237
- See also: Link to Prescribing Information — http://www.astellas.us/docs/amevive.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Started | 49 | 49
Completed Treatment | 42 | 44
Completed | 33 (Represents patients who completed follow-up) | 26 (Represents patients who completed follow-up)
Not Completed | 16 | 23
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 6 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 7 | 16
Not completed — Lack of Compliance | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alefacept Alone | Alefacept + nbUVB | Total
Number analyzed (Participants) | 49 | 49 | 98
Age Continuous [Mean (Standard Deviation); unit: years] | 48.2 (13.8) | 47.1 (14.2) | 47.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 37 | 32 | 69
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5 | 6 | 11
  Black | 0 | 1 | 1
  Caucasian | 43 | 42 | 85
  Other | 1 | 0 | 1
PGA Score [Mean (Standard Deviation); unit: Score] — The PGA scale is a tool used to evaluate the degree of overall lesion severity. The scale ranges from 0 (clear) to 5 (very severe).
  Score | 3.3 (0.7) | 3.4 (0.6) | 3.3 (0.6)
BSA Score [Mean (Standard Deviation); unit: Percentage of BSA] — The percentage of Body Surface Area (BSA) covered with Psoriasis.
  Percentage of BSA | 21.9 (13.0) | 20.0 (9.4) | 21.0 (11.3)
DLQI Score [Mean (Standard Deviation); unit: Score] — The DLQI questionnaire is intended to measure how much a subject's skin problem affects the subject's life. Subjects provide answers considering the past week. The scale of the DQLI ranges from 0 (best) to 30 (worst).
  Score | 6.1 (10) | 5.9 (7) | 6.1 (9)
PASI Score [Mean (Standard Deviation); unit: Score] — The PASI score is a tool that allows investigators to assign an objective number to the degree of severity of a person's psoriasis, and considers: redness, scaling and thickness. Values for PASI score range from 0 (least) to 72 (worst).
  Score | 17.8 (6.0) | 17.5 (5.2) | 17.7 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieve Psoriasis Area and Severity Index (PASI) 75 at Week 16
Description: The PASI score is a tool that allows investigators to assign an objective number to the degree of severity of a person's psoriasis, and considers: redness, scaling and thickness. Values for PASI score range from 0 (least) to 72 (worst).
  PASI 75 was defined as an improvement of at least 75% in PASI as compared to Baseline.
  The Last Observation Carry Forward (LOCF) method was used to impute missing data.
Time Frame: Week 16
Population: The number of participants analyzed per arm represents the ITT-Efficacy Population, which consisted of all subjects randomized into the study who received at least one dose of study drug (alefacept).
Measure: Number; unit: Percentage of Subjects
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 49 | 49
Percentage of Subjects | 22.4 | 44.9
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Test type: Superiority or Other; p = 0.032, Fisher Exact — No adjustments were made for multiple comparisons

2. Secondary Outcome: Percentage of Subjects Reaching PASI 75 Over the Entire Course of the Study
Description: as for outcome 1
Time Frame: Week 36
Population: The number of participants analyzed per arm represents the ITT-Efficacy Population, which consisted of all subjects randomized into the study who received at least one dose of study drug (alefacept).
  Only subjects who completed follow-up were included in this analysis.
Measure: Number; unit: Percentage of Subjects
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 49 | 49
Percentage of Subjects | 26.5 | 36.7
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Test type: Superiority or Other; p = 0.037, Wilcoxon (Mann-Whitney) — No adjustments were made to multiple comparisons

3. Secondary Outcome: Change in Body Surface Area (BSA) Covered With Psoriasis at Week 16
Description: A negative change from Baseline represents improvement.
  Change is calculated as Week 16- Baseline.
  The Last Observation Carry Forward (LOCF) method was used to impute missing data.
Time Frame: Baseline and Week 16
Population: The number of participants analyzed per arm represents the ITT-Efficacy Population, which consisted of all subjects randomized into the study who received at least one dose of study drug (alefacept).
  The number of participants per arm is consistent for all categories / rows of the data table.
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 49 | 49
Percentage of BSA
  Baseline | 21.9 (13.0) | 20.0 (9.4)
  Week 16 | 13.9 (10.8) | 6.6 (8.0)
  Change from Baseline | -8.0 (14.7) | -13.4 (9.2)
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Statistical Analysis applies to 'Change from Baseline'; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney) — No adjustments were made for multiple comparisons

4. Secondary Outcome: Change in Body Surface Area (BSA) Covered With Psoriasis Over the Entire Course of the Study
Description: A negative change from Baseline represents improvement.
  Change is calculated as Week 36- Baseline.
  The Last Observation Carry Forward (LOCF) method was used to impute missing data.
Time Frame: Baseline and Week 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 49 | 49
Percentage of BSA
  Baseline | 21.9 (13.0) | 20.0 (9.4)
  Week 36 | 14.4 (14.1) | 8.2 (8.8)
  Change from Baseline | -7.5 (14.7) | -11.9 (9.7)
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Statistical Analysis applies to 'Change from Baseline'; Test type: Superiority or Other; p = 0.382, ANOVA — Results were adjusted for use of concomitant psoriasis treatment

5. Secondary Outcome: Percentage of Subjects Who Achieved Physical Global Assessment (PGA) of Clear or Almost Clear at Week 16
Description: The PGA scale is a tool used to evaluate the degree of overall lesion severity. The scale ranges from 0 (clear) to 5 (very severe). Clear is defined as a score of 0; Almost Clear is defined as a score of 1.
  Subjects who achieved PGA of clear or almost clear at any visit during the study were assigned to the YES category for their respective groups.
  The Last Observation Carry Forward (LOCF) method was used to impute missing data.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 49 | 49
Percentage of Subjects
  PGA Clear or Almost Clear = Yes | 22.5 | 42.9
  PGA Clear or Almost Clear = No | 77.6 | 57.1
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Statistical Analysis applies to 'Clear or Almost Clear = Yes'; Test type: Superiority or Other; p = 0.052, Fisher Exact — No adjustments were made for multiple comparisons

6. Secondary Outcome: Percentage of Subjects Who Achieved Physical Global Assessment (PGA) of Clear or Almost Clear Over the Entire Course of the Study
Description: as for outcome 5
Time Frame: Week 36
Population: as for outcome 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 49 | 49
Percentage of Subjects
  PGA of Clear or Almost Clear = Yes | 34.7 | 59.2
  PGA of Clear or Almost Clear = No | 65.3 | 40.8
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Statistical Analysis applies to 'Clear or Almost Clear = Yes'; Test type: Superiority or Other; p = 0.026, Fisher Exact — No adjustments were made for multiple comparisons

7. Secondary Outcome: Percentage of Subjects Who Achieve PASI 90 at Week 16
Description: The PASI score is a tool that allows investigators to assign an objective number to the degree of severity of a person's psoriasis, and considers: redness, scaling and thickness. Values for PASI score range from 0 (least) to 72 (worst).
  PASI 90 was defined as an improvement of at least 90% in PASI as compared to Baseline.
  The Last Observation Carry Forward (LOCF) method was used to impute missing data.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: Percentage of Subjects
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 49 | 49
Percentage of Subjects
  PASI 90 = Yes | 8.2 | 20.4
  PASI 90 = No | 91.8 | 79.6
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Statistical Analysis applies to 'PASI 90 = Yes'; Test type: Superiority or Other; p = 0.147, Fisher Exact — No adjustments were made for multiple comparisons

8. Secondary Outcome: Time to Relapse
Description: The analysis only included subjects who achieved a 75% improvement in PASI and then relapsed.
  Relapse is defined by a loss of 50% of improvement in PASI.
Time Frame: Week 36
Population: The number of participants analyzed per arm represents the ITT-Efficacy Population, which consisted of all subjects randomized into the study who received at least one dose of study drug (alefacept).
  Only subjects who achieved a 75% improvement in PASI and then relapsed were included in the analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 2 | 2
Days | 98.0 (19.8) | 119.0 (29.7)
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Test type: Superiority or Other; p = 0.566, Log Rank — No adjustments were made for multiple comparisons

9. Secondary Outcome: Time for 50% Decrease in PASI
Description: The PASI score is a tool that allows investigators to assign an objective number to the degree of severity of a person's psoriasis, and considers: redness, scaling and thickness. Values for PASI score range from 0 (least) to 72 (worst).
  Only subjects who experienced 50% decrease in PASI were included in the analysis.
Time Frame: Week 36
Population: The number of participants analyzed per arm represents the ITT-Efficacy Population, which consisted of all subjects randomized into the study who received at least one dose of study drug (alefacept).
  Only subjects who experienced a 50% decrease in PASI were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 29 | 44
Days | 84.0 [57.0 to 112.0] | 56.0 [53.5 to 68.5]
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Test type: Superiority or Other; p = 0.001, Log Rank — No adjustments were made for multiple comparisons

10. Secondary Outcome: Time for a 75% Decrease in PASI
Description: The PASI score is a tool that allows investigators to assign an objective number to the degree of severity of a person's psoriasis, and considers: redness, scaling and thickness. Values for PASI score range from 0 (least) to 72 (worst).
  Only subjects who experienced 75% decrease in PASI were included in the analysis.
Time Frame: Week 36
Population: The number of participants analyzed per arm represents the ITT-Efficacy Population, which consisted of all subjects randomized into the study who received at least one dose of study drug (alefacept).
  Only subjects who experienced a 75% decrease in PASI were included in the analysis.
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 16 | 29
Days | 99.5 [83.0 to 135.0] | 84.0 [56.0 to 87.0]
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Test type: Superiority or Other; p = 0.007, Log Rank — No adjustments were made for multiple comparisons

11. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI)
Description: The DLQI questionnaire is intended to measure how much a subject's skin problem affects the subject's life. Subjects provide answers considering the past week. The scale of the DQLI ranges from 0 (best) to 30 (worst).
  A negative change from Baseline represents improvement.
  Change is calculated as Week 36- Baseline.
  The Last Observation Carry Forward (LOCF) method was used to impute missing data.
Time Frame: Baseline and Week 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: DLQI Score
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Number analyzed (Participants) | 49 | 49
DLQI Score
  Baseline | 11.0 (6.1) | 9.1 (5.9)
  Week 36 | 8.2 (7.6) | 5.6 (6.7)
  Change from Baseline | -2.7 (6.5) | -3.5 (6.4)
Statistical Analysis 1: Comparison: Alefacept Alone vs Alefacept + nbUVB; Statistical Analysis applies to 'Change from Baseline'; Test type: Superiority or Other; p = 0.539, ANOVA — Results were adjusted for use of concomitant psoriasis treatment

ADVERSE EVENTS:
Time Frame: From the time of Informed Consent through the last study visit.
Arm/Group | Alefacept Alone | Alefacept + nbUVB
Serious Adverse Events (participants affected / at risk) | 0/49 | 2/49
Other Adverse Events (participants affected / at risk) | 10/49 | 40/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alefacept Alone (N=49) | Alefacept + nbUVB (N=49)
Edema legs (General disorders) | 0 | 1
Cervical disc herniation (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical cord compression (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alefacept Alone (N=49) | Alefacept + nbUVB (N=49)
Common cold (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 6
CD4 lymphocytes decreased (Investigations) | 10 | 7
Erythema (Skin and subcutaneous tissue disorders) | 0 | 33
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 5

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.